CLINICAL TRIAL: NCT05049096
Title: Focused Power Ultrasound Mediated Inferior Perirenal Adipose Tissue Modification Therapy for Essential Hypertension: a Multicenter, Randomized, Double-blinded Controlled Trial. PARADISE Study
Brief Title: Focused Power Ultrasound Mediated Inferior Perirenal Adipose Tissue Modification Therapy for Essential Hypertension
Acronym: PARADISE-HTN
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Till interim analysis, 100 cases were enrolled, 71 of which during the COVID-19. Affected by epidemic control policy, 58 cases had examination window exceeded or missed, causing significant impact on endpoints, so we decided to terminate the trial.
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PARADISE-HTN
Record Dates: First submitted 2021-09-07; First posted 2021-09-17 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-12

CONDITIONS: Hypertension; Blood Pressure; Cardiovascular Diseases
Keywords: Hypertension; Cardiovascular disease; Focused ultrasound; Novel method
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: This is a ramdomized, double-blinded, and sham-control study. The ratio of the intervention group versus sham-control group is 1:1
Who Masked: Participant, Care Provider, Investigator
Masking Description: The masking range includes participants, most researchers (including the study leader; subjects screening researchers; follow-up researchers; sonographers; MR scanners, members of the clinical endpoint identification committee,and etc.) except for the study statistical analysts and the therapy operators
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): In intervention group, participants will receive the whole peri-renal fat modification therapy (including peri-renal fat ultrasonic measurement and localization,focused ultrasound treatment parameters setting and initiating)
  Interventions: Device: focused power ultrasound mediate inferior perirenal adipose tussue modification
- sham-control group (Sham Comparator): In sham control group, participants will receive the sham control therapy(including peri-renal fat ultrasonic measurement and localization,focused ultrasound treatment parameters setting),however,without initiating the focused ultrasound equipment.
  Interventions: Device: sham-control group

INTERVENTIONS:
Device: focused power ultrasound mediate inferior perirenal adipose tussue modification — This novel focused power ultrasound is an externally delivered, completely noninvasive focused therapeutic ultrasound device. It is capable of focusing the resulting ultrasound beam to a small "cigar"-shaped volume and monitoring the temperature of the target area, which leads to the rapid elevation of the peri-renal adipose tissue temperature and the destruction of target tissue eventually.
  Arms: intervention group
Device: sham-control group — participants will receive the sham control therapy(including peri-renal fat ultrasonic measurement and localization,focused ultrasound treatment parameters setting),however,without initiating the focused ultrasound equipment.
  Arms: sham-control group

SUMMARY:
This randomized, double blinded, sham-control trial aims to evaluate the efficacy and safety of a novel focused power ultrasound mediated inferior perirenal adipose tissue modification therapy for essential hypertension.

DETAILED DESCRIPTION:
The increase of visceral fat is closely related to the occurrence of hypertension, and it is one of the main independent risk factors of hypertension. Visceral fat has been recognized as an important endocrine organ, and a variety of factors secreted by visceral fat lead to an increased risk of cardiovascular disease. Peri-renal fat is a special type of visceral fat which is different from other type of visceral fat in histology, physiology, and functions. The positon of peri-renal fat is more stable than other visceral fat, which might be influenced by breath or body position changes.Studies have found that perirenal fat is an early predictor of ASCVD, and its accumulation is closely related to the occurrence and development of ASCVD.Therefore, the reduction or modification of visceral fat,especially peri-renal fat , has a sufficient scientific basis for the treatment of hypertension.

In our previous experiments, this novel focused power ultrasound can rapidly and efficiently promote the perirenal adipse tissue fibrosis and control the blood pressure in the model of swine. Moreover, we performed a single arm, small sample study to investigate the feasibility of the novel focused power ultrasound to modify the inferior perirenal adipose tissue in human volunteers, showing that this kind of method was feasible and safe.

In this study, we aim to further evaluate the efficacy and safety of a novel focused power ultrasound mediated inferior perirenal adipose tissue modification therapy for essential hypertension.

ELIGIBILITY:
Inclusion Criteria:

1. Individual has office systolic blood pressure (SBP) ≥ 140 mmHg and <180 mmHg when receiving a medication regimen of one, two, or three antihypertensive medication classes；
2. Individual has 24-hour Ambulatory Blood Pressure Monitoring (ABPM) average SBP≥135 mmHg；
3. The anteroposterior, transverse and axial diameters of inferior perirenal fat pad measured by ultrasound should be at least 20mm；
4. Individual is willing to sign the informed consent of the study.

Exclusion Criteria:

1. Individual is diagnosed as secondary hypertension (e.g. renal parenchymal hypertension, renal artery stenosis, primary aldosteronism, pheochromocytoma, Cushing's syndrome, aortic coarctation, obstructive sleep apnea hypopnea syndrome)；
2. Individual has history of kidney and or kidney surrounding tissue surgery;
3. Individuals has impairment of liver or kidney function (ALT, AST or creatinine is greater than 2 times of the upper limit of normal reference);
4. Individual has myocardial infarction, unstable angina pectoris, cerebrovascular accident or transient ischemic attack within 6 months of enrollment;
5. Individual has type 1 diabetes or poorly-controlled type 2 diabetes；
6. Individual has uncontrolled thyroid dysfunction;
7. Individual has urinary calculi and/or hematuria；
8. Individual has atrial fibrillation;
9. Individual has severe structural heart disease (e.g. heart valve disease, cardiomyopathy, congenital heart disease);
10. Individual has second degree and above atrioventricular block；
11. Individual has abnormal coagulation function;
12. Individual has infected waist skin;
13. Individual has malignant tumor;
14. Individual is pregnant, nursing or planning to be pregnant;
15. Individual is unwilling to sign informed consent;
16. Individual fails to complete the screening period.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2023-11-20 (Actual)

PRIMARY OUTCOMES:
Office Systolic Blood Pressure | From baseline to 1 month post-procedure
  Changes of office systolic blood pressure at 1-month compared with baseline

SECONDARY OUTCOMES:
Office Systolic Blood Pressure | From baseline to 3 months post-procedure
  Changes of office blood pressure at 3-month compared with baseline
Ambulatory Blood Pressure | From baseline to 1 month post-procedure
  Changes of mean systolic blood pressure measured by 24-hour ambulatory blood pressure monitoring at 1-month compared with baseline
Ambulatory Blood Pressure | From baseline to 3 months post-procedure
  Changes of mean systolic blood pressure measured by 24-hour ambulatory blood pressure monitoring at 3-month compared with baseline
Heart Rate | From baseline to 1 month post-procedure
  Changes of the heart rate at 1-month compared with baseline
Mean Heart Rate | From baseline to 1 month post-procedure
  Changes of the mean heart rate measured by 24-hour ambulatory blood pressure monitoring at 1-month compared with baseline

OTHER OUTCOMES:
Safety evaluation | From baseline to 1 month post-procedure
  Any severe adverse events (SAE) related to intervention. The SAE were defined as acute renal failure, acute intestinal perforation, and thromboembolic events, et al.

CONTACTS AND LOCATIONS:
Overall Officials: Xiangqing Kong, MD, Principal Investigator — Jiangsu province Hospital/The First Affiliated Hospital of Nanjing Medical University
Locations (3):
- China (3):
  - Jiangsu Province Hospital/The Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - The Affiliated Jiangning Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Suzhou Municipal Hospital, Suzhou, Jiangsu

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hayashi T, Boyko EJ, Leonetti DL, McNeely MJ, Newell-Morris L, Kahn SE, Fujimoto WY. Visceral adiposity is an independent predictor of incident hypertension in Japanese Americans. Ann Intern Med. 2004 Jun 15;140(12):992-1000. doi: 10.7326/0003-4819-140-12-200406150-00008. PMID 15197016
- [Result] Chandra A, Neeland IJ, Berry JD, Ayers CR, Rohatgi A, Das SR, Khera A, McGuire DK, de Lemos JA, Turer AT. The relationship of body mass and fat distribution with incident hypertension: observations from the Dallas Heart Study. J Am Coll Cardiol. 2014 Sep 9;64(10):997-1002. doi: 10.1016/j.jacc.2014.05.057. PMID 25190234
- [Result] Djawari D, Haneke E. [Therapy of recurrent oral aphthae with thymopoetin pentapeptide]. Hautarzt. 1983 Sep;34(9):463-4. German. PMID 6355012
- [Derived] Hua Y, Li MH, Lou YX, Zhang KR, Yang JM, Sheng YH, Zhang YQ, Cheng CL, Zou C, Wu TT, Kong XQ, Sun W. Perirenal fat as a potential marker and therapeutic target for metabolic syndrome: insights from a multicenter randomized controlled trial. Front Endocrinol (Lausanne). 2025 May 23;16:1557701. doi: 10.3389/fendo.2025.1557701. eCollection 2025. PMID 40487756
- [Derived] Li M, Shi J, Sheng Y, Zhang Y, Wu T, Yang J, Zhang K, Sun W, Kong X. Effect of focused power ultrasound-mediated perirenal fat modification on primary hypertension: protocol of a multicenter, randomized, double-blinded, sham-controlled study. Trials. 2023 Mar 23;24(1):221. doi: 10.1186/s13063-023-07249-5. PMID 36959658